CLINICAL TRIAL: NCT06960486
Title: Bedside Ultrasound-guided Real-time Biliary Drainage by Emergency Surgeon Improving Prognosis in the Frail and High Risk Elderly Patients With Severe Acute Suppurative Infection of Biliary Tract: A Randomised Controlled Trial
Brief Title: Ultrasound-guided Biliary Drainage Improving Prognosis in the Frail and High Risk Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Chunjie Liu, professor, Hebei Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180063
Record Dates: First submitted 2025-04-09; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Biliary Tract Infection
Keywords: infection of biliary tract; emergency bedside ultrasound; ultrasound-guided biliary drainage
MeSH Terms: conditions — Cholangitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- emergency bedside ultrasound group (Experimental): The experimental group will be performed gallbladder or bile duct puncture under the guidance of emergency bedside ultrasound.
  Interventions: Procedure: Bedside ultrasound-guided real-time biliary drainage
- traditional ultrasound group (Other): The control group will be performed puncture by traditional appointment ultrasound.
  Interventions: Procedure: traditional appointment ultrasound

INTERVENTIONS:
Procedure: Bedside ultrasound-guided real-time biliary drainage — Bedside ultrasound-guided real-time biliary drainage by emergency surgeon in the frail and high risk elderly patients with severe acute suppurative infection of biliary tract
  Arms: emergency bedside ultrasound group
Procedure: traditional appointment ultrasound — Traditional appointment ultrasound
  Arms: traditional ultrasound group

SUMMARY:
Acute biliary tract infection is a kind of disease caused by bacteria of biliary tract infection, mainly including acute cholecystitis and acute cholangitis, especially acute obstructive suppurative cholangitis (AOSC),which can lead to septic shock and multiple organ failure,and the mortality rate is high in the frail and high risk elderly patients. Our study involved bedside ultrasoundguided real-time biliary drainage by emergency surgeon in the frail and high risk elderly patients with severe acute suppurative infection of biliary tract,the goal of this clinical trial is to learn if it can improve patient prognosis and reduce mortality.

Participants will be divided into experimental group (emergency bedside ultrasound group) and controlgroup (traditional ultrasound group). The experimental group will be performed gallbladder or bile duct puncture under the guidance of emergency bedside ultrasound, while the control group will be performed puncture by traditional appointment ultrasound, The accuracy of ultrasound diagnosis, the total time of examination and puncture treatment,complications, hospitalization time and expenses will be compared between the two groups.

DETAILED DESCRIPTION:
After admission, vital signs will be collected by nurses and scored according to the Canadian health and aging clinical frailty scale 3 . Emergency surgeons will evaluate patients' airway, respiratory and circulatory status and intervene according to their condition. For patients with stable vital signs, CT will be performed first. Patients with untable vital signs and hemodynamics, bedside ultrasound will be performed by an emergency surgeon while aggressive rescue measures and further CT scans will be performed if the patient's condition permitted.The patients in the experimental group will be diagnosed by emergency surgeon using Philips CX50 portable ultrasound and treated by ultrasound-guided puncture and drainage at the first time, these included ultrasound-guided percutaneous transhepatic gallbladder drainage (PTGD) and percutaneous transhepatic choledochal drainage (PTCD) .In the control group, the patients will be scheduled for puncture and drainage treatment in the traditional ultrasound department at the same time of stabilizing vital signs.Then the two groups of patients will be followed up, through CT results to understand the accuracy of emergency bedside ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years.
* Patients with severe acute cholecystitis, and/or acute obstructive suppurative cholangitis who need emergency bedside ultrasound-guided biliary tract puncture.
* All patients were informed and volunteered to participate in the study.

Exclusion Criteria:

* Age < 75 years old.
* Patients who died before being admitted to the hospital for puncture treatment.
* Patients with severe bleeding tendency and coagulopathy.
* Patients who could not cooperate with the examination for any reason.
* Patients with a history of mental illness.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Puncture time | From admission time to completion of puncture time, assessed up to 3 hours
  Total time between admission and completion of ultrasound puncture
Hospitalization time | From hospitalization to discharge, about 30days
  hospitalization time
Hospitalization cost | From admission to the end of treatment, about 30 days
  Hospitalization expenses

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No